CLINICAL TRIAL: NCT06077955
Title: The Incidence of Gastrojejunostomy Ulceration After MGB-OAGB: Comparison of Hand-Sewn and Stapled Techniques of Anastomosis Formation. Multicenter Prospective Randomized Clinical Trial Study
Brief Title: Ulcers Formation After Hand-Sewn vs Stapled Gastrojejunal Anastomosis In MGB.
Acronym: ULTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Aleksandr E. Neimark, Leading researcher, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0210-22-MGB-OAGB
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Ulcer Peptic
Keywords: bariatric; morbid obesity; ulcer of gastrojejunostomy; mini-gastric bypass; one-anastomosis gastric bypass; hand-sewn anastomosis; stapled anastomosis
MeSH Terms: conditions — Peptic Ulcer; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Two groups: group A, a variant of the surgery with the stapled formation of a GJS, and group B, a variant with a hand-sewn formation of a GJS.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control) - with stapled anastomosis (Active Comparator): A variant of the surgery with the stapled formation of a gastrojejunostomy.
  Interventions: Procedure: Mini-gastric bypass with stapled anastomosis
- Group B (study) - with hand-sewn anastomosis (Experimental): A variant with a hand-sewn formation of a gastrojejunostomy.
  Interventions: Procedure: Mini-gastric bypass with hand-sewn anastomosis

INTERVENTIONS:
Procedure: Mini-gastric bypass with stapled anastomosis — the stomach is transected using linear endoscopic staplers in such a way as to create an isolated narrow gastric tube ("small ventricle") at least 17-18 cm long and 15-20 mm wide (diameter of gastric tube used 36-39 Fr). • A gastroenterostomy is performed at a distance of 150-200 cm from the ligament of Treitz using a linear stapler.
  Arms: Group A (control) - with stapled anastomosis
Procedure: Mini-gastric bypass with hand-sewn anastomosis — the stomach is transected using linear endoscopic staplers in such a way as to create an isolated narrow gastric tube ("small ventricle") at least 17-18 cm long and 15-20 mm wide (diameter of gastric tube used 36-39 Fr). • A gastroenterostomy is performed at a distance of 150-200 cm from the ligament of Treitz using a fully manual suture.
  Arms: Group B (study) - with hand-sewn anastomosis

SUMMARY:
We assume that the frequency of gastrojejunostomy ulcers after MGB-OAGB is associated with the peculiarities of the side-to-side gastrojejunostomy (GJS) formation, which is currently the "gold standard" for this procedure. The geometry of such anastomosis leads to the formation of a narrow strip of the gastric wall between two stapler lines (between the suture from the 2nd cassette during the formation of the "small ventricle" and directly from the suture from the cassette during the GJS formation). Perhaps this section of the stomach wall is prone to ischemia, which can certainly increase the risk of ulcer formation. It is also possible that a zone with impaired blood supply may also form in the "blind pocket" above the anastomosis.

When forming a Hand-Sewn GJS of the end-to-side type, ischemia zones do not occur. The anastomosis has a more physiological geometry, there is no conflict between the lines of stapled sutures.

Thus, we put forward the assumption that a serious risk factor for the development of a GJS ulcer was eliminated when switching to a completely manual technique for the GJS formation when performing MGB-OAGB.

The study is aimed at the compare the incidence of GJS ulcers during MGB-OAGB, depending on the techniques of anastomosis formation.

DETAILED DESCRIPTION:
Today, MGB-OAGB, a mini-gastric bypass or one anastomosis gastric bypass, is one of the most widely used bariatric procedures. This surgery was first performed by Professor R. Rutledge in 1997, having published the first data in 2001 on a sample of 1274 patients [1]. In 2014, the first consensus conference was held, at which recommendations for application and generalization of experience were adopted [2]. By 2018, the share of MGB-OAGB surgeries in the world was already 7.7% [3]. In the Russian Federation, this index for 2021 was 12%, which indicates a significant prevalence of mini-gastric bypass surgery in the Russian Federation [4]. This is facilitated by the simplicity, safety and high efficiency of this procedure in relation to obesity and metabolic disorders. Comparative studies and subsequent meta-analyses show a number of advantages over the classic Roux-en-Y gastric bypass [5, 6]. Reduction in the duration of the surgery and the reduction in the number of surgical complications are attractive for surgeons.

However, with the increase in the number of surgeries and the accumulation of experience, a number of problems associated with this surgery become apparent. Malabsorption risks are minimized by measuring the length of the common loop and cutting off a strictly defined percentage of the small intestine from digestion. Research on bile reflux effects is currently ongoing, but in order to reduce it, the surgical technique has been modified by lengthening the gastric tube [2]. One of the most serious problems is the appearance of gastrojejunostomy (GJS) ulcers. As a rule, they are difficult to treat and can cause bleeding. Their number seriously varies in different publications from 2% to 13% [7, 8]. These figures, despite the attractiveness of the new surgery, make many surgeons refrain from performing MGB-OAGB in their routine practice. The causes of ulcers are not fully understood and require further study, and it is also possible to change the technique of anastomosis.

Working Hypothesis We assume that the frequency of gastrojejunostomy ulcers after MGB-OAGB is associated with the peculiarities of the side-to-side GJS formation, which is currently the "gold standard" for this procedure. The geometry of such anastomosis leads to the formation of a narrow strip of the gastric wall between two stapler lines (between the suture from the 2nd cassette during the formation of the "small ventricle" and directly from the suture from the cassette during the GJS formation). Perhaps this section of the stomach wall is prone to ischemia, which can certainly increase the risk of ulcer formation. It is also possible that a zone with impaired blood supply may also form in the "blind pocket" above the anastomosis.

When forming a Hand-sewn GJS of the end-to-side type, ischemia zones do not occur. The anastomosis has a more physiological geometry, there is no conflict between the lines of stapled sutures.

Thus, we put forward the assumption that a serious risk factor for the development of a GJS ulcer was eliminated when switching to a completely Hand-sewn technique for the GJS formation when performing MGB-OAGB.

Purpose of the Study To compare the incidence of GJS ulcers during MGB-OAGB, depending on the techniques of anastomosis formation.

Materials and Research Methods In order to assess the target parameter and the endpoint of the study, all patients who underwent surgical treatment will undergo a video endoscopy of the upper gastrointestinal tract 6 months after surgical treatment.

As research tools, it is planned to use instrumental, laboratory and surgery equipment, as well as all other necessary material and technical equipment of the above medical institutions.

Treatment Protocol All eligible and randomized patients will undergo laparoscopic MGB-OAGB no later than 1 month after randomization and enrollment. As part of a standardized preoperative assessment, a set of examinations will be performed, see Appendix 2.

Standardized surgery protocol:

* One-time antibacterial prophylaxis is performed, activities are carried out for the induction of anesthesia, tracheal intubation and the implementation of inhalation anesthesia with mechanical ventilation in accordance with the local standards of the participating centers.
* Patient is placed in the supine position with the head of the bed elevated at 30° (Fowler's position).
* A carboxyperitoneum is created with a pressure of 12-16 mm Hg.
* Five trocars are installed in the upper mesogastrium according to the accepted technique for performing surgical interventions on the upper floor of the abdominal cavity in each specific clinical center.
* By one of the types of surgical energy (ultrasound, bipolar, monopolar) along the lesser curvature of the stomach, the lesser omentum is dissected and the omentum is entered from the omental bag at or distal to the crow's foot, the minimally necessary retrogastric adhesiolysis is performed.
* The gastroesophageal junction and the angle of His are mobilized. Then the stomach is transected using linear endoscopic staplers in such a way as to create an isolated narrow gastric tube ("small ventricle") at least 17-18 cm long and 15-20 mm wide (diameter of gastric tube used 36-39 Fr). Blue, green, gold, purple, and black cassettes (cassettes or cartridges in blue, green, black, or purple) can be used.
* Staple line hemostasis by applying clips.
* The greater omentum may be transversely incised depending on individual anatomy.
* Visualization of the ligament of Treitz.
* Measurement of the length of the small intestine at a distance of at least 5 m.
* A gastroenterostomy is performed at a distance of 150-200 cm from the ligament of Treitz using a linear stapler in group A and using a fully Hand-sewn suture in group B.
* Gastrotomy at the end section of the stapler line of the distal "small ventricle" and enterotomy at 150-200 cm from the ligament of Treitz are performed in group A. GJS is formed using a blue or purple cartridge (the height of the braces is 3.5 mm). The width of the formed anastomosis is calibrated according to the branch of the apparatus of 35-40 cm. The technological hole is closed with absorbable monofilament suture material with a biodegradation time of not more than 180 days on a pricking needle.
* Extended gastrotomy by cutting off the end stapler line (1st cassette, when forming the "small ventricle") is performed in group B. Enterotomy with a length of 35-40 mm is performed at a distance of 150-200 cm from the ligament of Treitz. GJS is formed by a manual single-row continuous suture using any absorbable monofilament suture material with a biodegradation period of not more than 180 days on a pricking needle.
* Performing an anastomosis leak test with a solution of methylene blue or bubble leak test.
* Testing for hemostasis.
* Desufflation of gas and suturing of trocar wounds are carried out.

After the surgical intervention, if necessary, the patient can be in the intensive care unit and monitoring until the stabilization of the condition, then transferred to the specialized surgical department.

Recommendations for nutrition after surgery: oral intake of light glucose-containing liquids begins on the first postoperative day (6-12 hours after surgery). On the second day after the surgery, the intake of concentrated glucose-containing and complex nutritional drinks begins.

After discharge from the hospital, the patient must adhere to the protocol diet (Appendix 3). All patients will be required to take preventive therapy with an established PPIs 40 mg daily for 6 months after surgery.

Intermediate Control From the moment of discharge from the hospital until the moment of assessment of the target parameter, remote monitoring will be carried out to control the patient's compliance (regularity of PPI intake, adherence to recommendations on the postoperative diet) and complaints, possibly associated with the early onset of erosive and ulcerative lesions of the upper gastrointestinal tract. Telephone control will be carried out in periods of 1, 2, 3 and 5 months after surgical treatment.

In the event of a premature referral of the patient or detection of complaints during the intermediate control, indicating the possible development of erosive and ulcerative lesions of the upper gastrointestinal tract, the patient will undergo a premature flexible endoscopy of the upper gastrointestinal tract. If a GJS ulcer is detected, the endpoint will prematurely be assessed as positive.

Expected Results It is expected to reveal a statistically significant reduction in the incidence of GJS ulceration when performing MGB-OAGB using a Hand-sewn anastomosis technique compared with a stapled technique.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65;
* Body mass index over 40 kg/m2 or 35 kg/m2 in the presence of concomitant metabolic disorders (type 2 diabetes mellitus, hypertension, coronary artery disease, atherosclerosis and dyslipidemia);
* Preliminary consultation with an endocrinologist;
* Voluntary informed consent for surgical treatment;
* Voluntary informed consent to participate in a clinical trial;
* A negative test for Helicobacter pylori or a full course of eradication therapy.

Non-Inclusion Criteria:

* smoking;
* gastric ulcer disease in history;
* earlier abdominal surgery by laparotomy
* abdominal wall hernias;
* contraindications to planned operative treatment of bariatric profile based on the results of the pre-surgery evaluation of somatic status (see section "Patient's Treatment Protocol");
* for women - pregnancy planning in the next 12 months;
* mental health record;
* patients with oncological diseases;

Exclusion Criteria:

* surgical complications in the early post-surgery period related to the disruption of vital functions of organs and systems (respiratory, neurological and cardiological disorders requiring a stay in then the intensive-care unit, long-term position compression syndrome with renal impairment, venous thromboembolism);
* surgical complications in the early post-surgery period requiring repeated surgery or minimally invasive surgery (intraabdominal / intraluminal hemorrhage, failure of manual/ hardware suture on gastrointestinal organs etc.);
* positive intraoperative test for leak-proof anastomosis (injection of methylene blue solution or "bubble-test"), requiring surgical procedures for color leakage zone removal (see section "Patient's Treatment Protocol");
* poor adherence to the recommendations for gastroprotective therapy and recommendations on diet after surgery by the patient (see section "Interim control");
* patient's refusal to participate in the clinical study at any stage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The presence of a gastrojejunostomy ulcer | 6 months
  Video endoscopy of the upper gastrointestinal tract

SECONDARY OUTCOMES:
Erosive anastomositis | 6 months
  Video endoscopy of the upper gastrointestinal tract
Time of surgery | Intraoperative indicator
  Operation time from skin incision to completion of skin suturing
The amount of foreign non-absorbable material remaining in the body | Intraoperative indicator
  The number of cartridges from staplers used during the operation is counted

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Neimark, MD, PhD, Principal Investigator — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutledge R. The mini-gastric bypass: experience with the first 1,274 cases. Obes Surg. 2001 Jun;11(3):276-80. doi: 10.1381/096089201321336584. PMID 11433900
- [Background] Ramos AC, Chevallier JM, Mahawar K, Brown W, Kow L, White KP, Shikora S; IFSO Consensus Conference Contributors. IFSO (International Federation for Surgery of Obesity and Metabolic Disorders) Consensus Conference Statement on One-Anastomosis Gastric Bypass (OAGB-MGB): Results of a Modified Delphi Study. Obes Surg. 2020 May;30(5):1625-1634. doi: 10.1007/s11695-020-04519-y. PMID 32152841
- [Background] Welbourn R, Hollyman M, Kinsman R, Dixon J, Liem R, Ottosson J, Ramos A, Vage V, Al-Sabah S, Brown W, Cohen R, Walton P, Himpens J. Bariatric Surgery Worldwide: Baseline Demographic Description and One-Year Outcomes from the Fourth IFSO Global Registry Report 2018. Obes Surg. 2019 Mar;29(3):782-795. doi: 10.1007/s11695-018-3593-1. Epub 2018 Nov 12. PMID 30421326
- [Background] National Bariatric Registry. URL: https://bareoreg.ru (Accessed: 01.08.2023).
- [Background] Ruiz-Tovar J, Carbajo MA, Jimenez JM, Castro MJ, Gonzalez G, Ortiz-de-Solorzano J, Zubiaga L. Long-term follow-up after sleeve gastrectomy versus Roux-en-Y gastric bypass versus one-anastomosis gastric bypass: a prospective randomized comparative study of weight loss and remission of comorbidities. Surg Endosc. 2019 Feb;33(2):401-410. doi: 10.1007/s00464-018-6307-9. Epub 2018 Jun 25. PMID 29943058 (Retraction: PMID 33452565 Surg Endosc. 2021 Mar;35(3):1492)
- [Background] Wang FG, Yan WM, Yan M, Song MM. Outcomes of Mini vs Roux-en-Y gastric bypass: A meta-analysis and systematic review. Int J Surg. 2018 Aug;56:7-14. doi: 10.1016/j.ijsu.2018.05.009. Epub 2018 May 16. PMID 29753952
- [Background] Mahawar KK, Reed AN, Graham YNH. Marginal ulcers after one anastomosis (mini) gastric bypass: a survey of surgeons. Clin Obes. 2017 Jun;7(3):151-156. doi: 10.1111/cob.12186. Epub 2017 Mar 20. PMID 28320077
- [Background] Baksi A, Kamtam DNH, Aggarwal S, Ahuja V, Kashyap L, Shende DR. Should Surveillance Endoscopy Be Routine After One Anastomosis Gastric Bypass to Detect Marginal Ulcers: Initial Outcomes in a Tertiary Referral Centre. Obes Surg. 2020 Dec;30(12):4974-4980. doi: 10.1007/s11695-020-04864-y. Epub 2020 Jul 27. PMID 32720263